CLINICAL TRIAL: NCT01177345
Title: Survey Assessment and Projection of the Social and Economic Burdens of Cervical Cancer in Tanzania
Brief Title: Burden of Cervical Cancer in Tanzania
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Olola Oneko, Kilimanjaro Christian Medical Centre, Tanzania
Other Study IDs: 36813
Record Dates: First submitted 2010-07-27; First posted 2010-08-09 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Cervical Cancer; -Socioeconomic Burden of Disease
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Terminal Disease: Terminal cervical cancer- not treatable
- Early Disease: Early cervical cancer = meaning treatable with hysterectomy.
- Advanced Disease: Advanced cervical cancer- treatable with chemotherapy and/or radiation.

SUMMARY:
Cervical cancer screening is a worldwide problem especially in the developing world of which Tanzania belongs. It is diagnosed late in the third world because there are no diagnostic facilities and resource people. It occurs in the age groups between 40 and above and therefore affects the productive age of the community. It is well known that women generally are the backbone of every community and specifically in the developing countries.

The objective of this research is to analyze and quantify the burden of cervical cancer disease in the community. It will research the interpersonal and socioeconomic issues associated with cervical cancer disease in the family.

ELIGIBILITY:
Inclusion Criteria:

* new pathological diagnosis of cervical cancer

Exclusion Criteria:

* non consenting individuals

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with cervical cancer at the Reproductive Health Clinic at Kilimanjaro Christian Medical Centre (KCMC) and satellite cervical cancer screening clinics in rural areas affiliated with KCMC.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Socioeconomic burden to households | 12 months
  1. share of household consumption attributable to medical care (hospitals, dispensaries, etc.)
  2. monthly household income (work hours, income sources, changes in the type or amount)
  3. child school attendance, nutrition (school days missed in past week, meals eaten, source of proteins on day prior to interview)

SECONDARY OUTCOMES:
Projection of economic impact on community | 12 months
  Combine rates of cervical cancer with the age and gender distribution in the Kilimanjaro Region (Tanzania Census), distribution of cancer stages, and primary outcomes from the study cohort to estimate of total medical expenses, income losses, and school days missed due to cervical cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Kilimanjaro Christian Medical Center, Moshi, Kilimanjaro, Tanzania